CLINICAL TRIAL: NCT01499719
Title: Surgery Checklist and Process Improvement Surrounding Endoscopic Sinus Surgery
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Dr. Timothy L. Smith, Principal Investigator, Oregon Health and Science University
Other Study IDs: checklist pause
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Rhinosinusitis
Keywords: Sinusitis; Disease; Chronic; Sinonasal
MeSH Terms: conditions — Sinusitis; Disease; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical checklist: Compliance for surgical checklist
  Interventions: Behavioral: Checklist introduction / Pause

INTERVENTIONS:
Behavioral: Checklist introduction / Pause — Operating room staff will be introduced to a new checklist specifically designed to address concerns around protocols for endoscopic sinus surgery to raise awareness and attention to 11 specific areas of interest.

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness of a new surgical checklist in the setting of sinus surgery for patients with chronic rhinosinusitis (CRS) and to measure the frequency of compliance by surgical personnel at OHSU with specific daily safety protocols before and after introduction of the checklist. The investigators hypothesized that the use of an ESS specific surgical checklist will improve the frequency of compliance by surgical personnel at OHSU to internal safety concerns and protocols.

DETAILED DESCRIPTION:
A total of 200 unidentified, non-randomized endoscopic sinus surgery cases will be observed and reviewed by research personnel (T.L.S, J.C.) within the Oregon Sinus Center, located within the Center for Health and Healing on the South Waterfront Campus of OHSU, under the direction of Timothy L. Smith, MD, MPH (PI). The first 100 surgical cases will be evaluated as "pre-intervention" cases by research personnel while the second 100 surgical cases will be evaluated as "post-intervention" cases after the introduction and discussion of the surgical checklist to operating room staff.

ELIGIBILITY:
Inclusion Criteria:

* CRS defined by 2007 Adult Sinusitis Guidelines.13
* Unidentified adult patients electing endoscopic sinus surgery for the treatment of CRS.

Exclusion Criteria:

* Unable to complete surgical procedures due to perioperative complications.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Resident and fellow surgeons.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sinus surgery checklist | 6 months
  11 dichotomous questions regarding observed operating room protocols for internal process improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States